CLINICAL TRIAL: NCT02651142
Title: Sentinel Lymph Node Biopsy With or Without Para-Sentinel Lymph Node Dissection in Breast Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Qifeng Yang, Chairman of Department of Breast Surgery, Qilu Hospital, Shandong University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HECT003
Record Dates: First submitted 2016-01-07; First posted 2016-01-08 (Estimated); Last update posted 2020-06-02 (Actual); Status verified 2020-05

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- SLNB with para-SLN dissection (Experimental): patients receive sentinel lymph node biopsy patients receive para-sentinel lymph node dissection
  Interventions: Procedure: Patients receive SLNB
- SLNB without para-SLN dissection (Experimental): patients received sentinel lymph node biopsy
  Interventions: Procedure: Patients receive SLNB

INTERVENTIONS:
Procedure: Patients receive SLNB — Patients receive sentinel lymph node biopsy

SUMMARY:
Sentinel lymph node biopsy（SLNB） is an established way of predicting axillary nodal metastasis in early breast cancer. We aim to determinethe，in a prospective randomized, controlled trial, effect of sentinel lymph node biopsy with para-sentinel lymph node(SLN) dissection versus sentinel lymph node biopsy without para-sentinel lymph node dissection on outcomes after breast surgery.

DETAILED DESCRIPTION:
Aim: Compare the disease-free survival (DFS) and overall survival (OS) of breast cancer patients who are randomized to receive sentinel lymph node biopsy with para-sentinel lymph node dissection group vs. those receive only sentinel lymph node biopsy without para-sentinel lymph node dissection

Outline:

Patients are randomized assigned to the following one of two groups and are followed annually.

Arm I: Patients receive sentinel lymph node biopsy with para-sentinel lymph node dissection Arm II: Patients receive only sentinel lymph node biopsy without para-sentinel lymph node dissection

ELIGIBILITY:
Inclusion Criteria:

1. histologically confirmed primary breast cancer by core needle biopsy or excisional biopsy
2. abnormal para-sentinel lymph node was found by ultrasound examination
3. ultrasound-guided fine needle aspiration cytology of these nodes were performed
4. the result of fine needle aspiration cytology was negative (no tumour cell was found)
5. patient planed to perform SLNB

Exclusion Criteria:

1. pathological diagnosed ductal carcinoma in situ by excisional biopsy
2. the result of fine needle aspiration cytology was positive
3. patient has received neo-adjuvant system therapy

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2015-01; Primary Completion 2021-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Disease free survival | Up to 10 years
  Time from randomization to recurrence, metastasis, appearance of a second primary tumor, or death from any cause, whichever occurs first, assessed up to 10 years.

SECONDARY OUTCOMES:
Overall survival | Up to 10 years
  Time from randomization to death from any cause, assessed up to 10 years.

CONTACTS AND LOCATIONS:
Locations (1):
- Qifeng Yang, Jinan, Shandong, China

REFERENCES:
- [Derived] Ma X, Wen S, Liu B, Li D, Wang X, Kong X, Ma T, Jiang L, Yang Q. Relationship between Upper Extremity Lymphatic Drainage and Sentinel Lymph Nodes in Patients with Breast Cancer. J Oncol. 2019 Apr 1;2019:8637895. doi: 10.1155/2019/8637895. eCollection 2019. PMID 31057616
- [Derived] Li X, Chen S, Jiang L, Kong X, Ma T, Xu H, Yang Q. Precise intraoperative sentinel lymph node biopsies guided by lymphatic drainage in breast cancer. Oncotarget. 2017 Jun 27;8(38):63064-63072. doi: 10.18632/oncotarget.18624. eCollection 2017 Sep 8. PMID 28968971